CLINICAL TRIAL: NCT05019001
Title: A Prospective Study Comparing the Efficacy of Laminoplasty and Laminectomy With Fusion for Ossification of the Posterior Longitudinal Ligament With High Occupation Rate in Cervical Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChenxinPekingUTH
Record Dates: First submitted 2021-06-20; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-06

CONDITIONS: Ossification of the Posterior Longitudinal Ligament
Keywords: OPLL; high occupation rate; laminoplasty; laminectomy with fusion
MeSH Terms: conditions — Ossification of Posterior Longitudinal Ligament | interventions — Laminoplasty; Laminectomy; Gene Fusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laminoplasty (Other): A posterior approach surgical method to treat patients with Ossification of the Posterior Longitudinal Ligament
  Interventions: Procedure: Laminoplasty
- Laminectomy With Fusion (Other): Another posterior approach surgical method to treat patients with Ossification of the Posterior Longitudinal Ligament
  Interventions: Procedure: Laminectomy With Fusion

INTERVENTIONS:
Procedure: Laminoplasty — A posterior approach surgical method to treat patients with Ossification of the Posterior Longitudinal Ligament
  Arms: Laminoplasty
Procedure: Laminectomy With Fusion — Another posterior approach surgical method to treat patients with Ossification of the Posterior Longitudinal Ligament
  Arms: Laminectomy With Fusion

SUMMARY:
The efficacy of laminoplasty and laminectomy with fusion for ossification of the posterior longitudinal ligament with high occupation rate in the cervical spine is not clear in the literature report so far. This study is designed to further research the difference in efficacy between the two surgical methods.

DETAILED DESCRIPTION:
Ossification of the posterior longitudinal ligament(OPLL) is a common spinal disease which can lead to neurological dysfunction and its morbidity is related to genetic factors. OPLL is usually found in cervical spine and characterized by hypertrophy and ossification of the posterior longitudinal ligament in the rear of the corresponding cervical vertebral body, which can encroach the space in the spinal canal and compress the spinal cord and/or nerve roots of the corresponding segments, resulting in sensory and motor disorders of the limbs as well as visceral autonomic nervous dysfunction, leading to neurological dysfunction and even high paraplegia. It not only causes great harm but also brings heavy economic and spiritual burden to patients and society.

Although the surgical treatments for OPLL include anterior and posterior approach, the anterior approach requires excellent equipment and rich operation experience for surgery doctor. Many articles showed significantly higher complications rate in anterior approach than that of posterior approach. Posterior approach surgery is considered to be one of the effective treatment methods for OPLL in cervical spine. In the posterior approach, there are two commonly recognized surgical procedures, laminoplasty and laminectomy with fusion. The efficacy of laminoplasty and laminectomy with fusion for ossification of the posterior longitudinal ligament with high occupation rate in the cervical spine is not clear in the literature report so far. This study is designed to further research the difference in efficacy between the two surgical methods. The purpose of this study is to make patients get the biggest medical benefits and to make a right surgical treatment strategy when doctors treating patients with high occupation rate OPLL in cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed by clinical symptoms, physical examination, X-ray, CT, and MRI with a high occupation rate of ossification of the posterior longitudinal ligament in the cervical spine need and can be treated surgically after preoperative examination.
* CT axial soft tissue window determine that the occupation rate of one or more spinal canal segments in C2-7 is more than 60%.
* Sagittal CT show ossification of more than 3 segments of the posterior longitudinal ligament of the cervical spine.
* Sign the written informed consent

Exclusion Criteria:

* Participating in other interventional clinical trials;
* Mental disorders or cognitive disorders;
* Heart and lung diseases;
* Nervous system diseases;
* Patients with serious liver and kidney diseases, tumors and infectious diseases;
* There are any other factors that the treated doctors consider unsuitable for inclusion or completion of the study.
* Patients with cervical spondylotic radiculopathy
* Patients with severe osteoporosis, skeletal fluorosis and other reasons for which laminoplasty is not feasible
* Patients with ossification of posterior longitudinal ligament of cervical spine with invasion rate ≥60% had cervical trauma
* The patient with cervical ligamentum flavum ossification was diagnosed at the C2-7 level
* Preoperative pregnancy test was performed to exclude pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
preoperative mJOA score | preoperative
  Preoperative mJOA score, range from 0 to 17. The higher the score, the less severe the symptoms
postoperative mJOA score | postoperative at 3 months
  Postoperative mJOA score, range from 0 to 17. The higher the score, the less severe the symptoms
postoperative mJOA score | postoperative at 6 months
  Postoperative mJOA score, range from 0 to 17. The higher the score, the less severe the symptoms
postoperative mJOA score | postoperative at 1 year
  Postoperative mJOA score, range from 0 to 17. The higher the score, the less severe the symptoms
postoperative mJOA score | postoperative at 2 year
  Postoperative mJOA score, range from 0 to 17. The higher the score, the less severe the symptoms
mJOA score change rate | 3 months after surgery
  (Postoperative mJOA score-Preoperative mJOA score)/(17-Preoperative mJOA score)×100%
mJOA score change rate | 6 months after surgery
  (Postoperative mJOA score-Preoperative mJOA score)/(17-Preoperative mJOA score)×100%
mJOA score change rate | 1 year after surgery
  (Postoperative mJOA score-Preoperative mJOA score)/(17-Preoperative mJOA score)×100%
mJOA score change rate | 2 years after surgery
  (Postoperative mJOA score-Preoperative mJOA score)/(17-Preoperative mJOA score)×100%

SECONDARY OUTCOMES:
Operation time | during operation
  Operation time during operation
blood loss | during operation
  blood loss during operation, parameter is milliliter, which is caculated by anesthetist during operation
Rate of C5 nerve root palsy | C5 nerve palsy after operation immediately
  Whether patient has deltoid muscle strength decrease after operation. If there is, it means to appear C5 palsy.
hematoma incidence | hematoma after operation immediately
  hematoma after operation
Rate of spinal cord injury | spinal cord injury after operation immediately
  Whether patient has spinal cord injury after operation. If there is, it means to appear sensory and motor impairments of limbs and trunk.
range of motion | preoperation
  the movement range of cervical
range of motion | 3 months after surgery
  the movement range of cervical
range of motion | 6 months after surgery
  the movement range of cervical
range of motion | 1 year after surgery
  the movement range of cervical
range of motion | 2 years after surgery
  the movement range of cervical
neck pain VAS score | 3 months after surgery
  Visual Analog Score for pain of neck, range from 0-10, a higher score means more pain
neck pain VAS score | 6 months after surgery
  Visual Analog Score for pain of neck, range from 0-10, a higher score means more pain
neck pain VAS score | 1 year after surgery
  Visual Analog Score for pain of neck, range from 0-10, a higher score means more pain
neck pain VAS score | 2 years after surgery
  Visual Analog Score for pain of neck, range from 0-10, a higher score means more pain

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided